CLINICAL TRIAL: NCT06883487
Title: Exploratory Study on HER2 Detection Method and Positive Threshold for High-grade Serous Adenocarcinoma of the Ovary
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jing Li, vice-professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-259-01
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-04

CONDITIONS: Exploring HER2 Positive Diagnostic Criteria in High-grade Serous Ovarian Cancer; Observing the Effectiveness of Targeted HER2 ADC Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Specimen with the diagnosis of high-grade serous ovarian adenocarcinoma within 5 years. The International Federation of Gynecology and Obstetrics(FIGO) stage is II or above with complete follow-up data.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study without intervention

SUMMARY:
Ovarian cancer is the most lethal gynecological malignancy, and 70% of ovarian cancer patients are diagnosed late at the time of new diagnosis. Even after systematic treatment, 75% of patients still relapse within 3 years and 70% die within 5 years. The survival prognosis of platinum resistant and refractory ovarian cancer populations is currently an urgent issue that needs attention. Antibody drug conjugate (ADC) targeting human epidermal growth factor receptor 2 (HER2) significantly improved the survival prognosis of patients with multiple solid tumors, such as breast cancer, gastric cancer, colorectal cancer, etc. Anti HER2 drugs have been a research hotspot in the treatment of advanced ovarian cancer in recent years. The expression status of HER2 has a decisive impact on the efficacy of ADC drugs targeting HER2. However, there is still a lack of large-scale data on HER2 expression rate in ovarian cancer patients, and there is no clear detection standard to guide clinical practice, which restricts the application of anti-HER2 ADC drugs in ovarian cancer.

To address this critical clinical issue, we initiated this study, which was divided into two parts: ① Retrospective study: Using the existing 144 samples of high-grade serous epithelial ovarian cancer(HGSOC) in our center, we used immunohistochemistry (IHC), DNA in situ hybridization (ISH), and second-generation sequencing (NGS) techniques to detect HER2 status, clarify the relationship between HER2 expression rate and patient survival outcomes, and preliminarily explore the best detection techniques and corresponding positive judgment thresholds for evaluating HER2 status in HGSOC; ② Real world observational study: To verify the predictive value of the positive judgment threshold determined in ① for efficacy in 20 ovarian cancer patients who received HER2 targeted ADC drugs due to platinum resistance/platinum refractory and no other effective treatment options in clinical practice. The aim of this project is to explore for the first time a reliable and feasible method for assessing the expression status of HER2 in patients with epithelial ovarian cancer, in order to provide a basis for subsequent evaluation of targeted HER2 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological type: high-grade serous adenocarcinoma of the ovary
2. Pathological slices stored within 5 years
3. FIGO stage II or above
4. Complete clinical and follow-up data

Exclusion Criteria:

1. Slice quality control failure
2. Incomplete follow-up data

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathological specimen stored by the department of pathology in Sun Yat-sen Memorial Hospital with a clinical diagnosis of FIGO stage II or above and complete survival data
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Exploratory study on HER 2 detection method and positive threshold for high-grade serous adenocarcinoma of the ovary | 2027-3-31
  Use multiple methods to detect the expression of HER 2 in HGSOC pathological specimens to find out the positive threshold of HGSOC patients then validate the threshold by observing the effectiveness of targeted HER2 ADC drugs in platinum resistant/refractory ovarian cancer patients in the real world

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China